CLINICAL TRIAL: NCT03365609
Title: A Comparison of Four Different Treatment Regimens as the First-line Treatment of Helicobacter Pylori in Chinese Children and Investigation of Resistance and Impact factors-a Multicenter Study
Brief Title: A Comparison of Four Different Treatment Regimens of Helicobacter Pylori in Chinese Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ying HUANG (Other)
Collaborators: Guangzhou Women and Children's Medical Center (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Beijing Children's Hospital (Other); Tang-Du Hospital (Other)
Responsible Party: Sponsor-Investigator, Ying HUANG, The director of gastroenterology of Children's Hospital of Fudan, Children's Hospital of Fudan University
Organization: Children's Hospital of Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPT2017
Record Dates: First submitted 2017-11-20; First posted 2017-12-07 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Helicobacter Infections
MeSH Terms: conditions — Helicobacter Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- T-group (Experimental): T-group(triple therapy)
  Interventions: Drug: triple therapy
- S-group (Experimental): S-group( sequential therapy)
  Interventions: Drug: sequential therapy
- B-group (Experimental): B-group( bismuth quadruple therapy )
  Interventions: Drug: bismuth quadruple therapy
- C-group (Experimental): C-group( concomitant therapy)
  Interventions: Drug: concomitant therapy

INTERVENTIONS:
Drug: triple therapy — Omeprazole+Amoxicillin+Clarithromycin
  Arms: T-group
Drug: sequential therapy — the first 7 days : Omeprazole+Amoxicillin, the last 7 days: Omeprazole+Clarithromycin+Metronidazole
  Arms: S-group
Drug: bismuth quadruple therapy — Omeprazole+Amoxicillin+Metronidazole+Colloidal Bismuth Subcitrate
  Arms: B-group
Drug: concomitant therapy — Omeprazole+Amoxicillin+Clarithromycin+Metronidazole
  Arms: C-group

SUMMARY:
With the resistance of Helicobacter pylori increasing, low and unsatisfactory eradication rate (64%) have been observed with standard triple therapy in European children. Which regimen is appropriate for Chinese children? There is no large scale, multi center studies in China about treatment, CYP2C19 gene polymorphism, resistance rate and resistance genotype. Investigators want to perform a research to compare four different treatment regimens（triple therapy, sequential therapy, bismuth quadruple therapy and concomitant therapy）as the first-line treatment of Helicobacter pylori in Chinese children and investigation of resistance, impact factors and changes of microbiota after the therapy. The results of the study will provide theoretical basis to make the new guideline of diagnosis and therapy of Helicobacter pylori in Chinese children. It advance instruct and norm the clinical practice for Chinese pediatrician to increase the cure rate of Helicobacter pylori and decrease the resistance.

DETAILED DESCRIPTION:
Eligible children were randomly divided into four groups: standard triple therapy, sequential therapy, bismuth quadruple therapy and concomitant therapy. The course of treatment is 14 days. The primary outcome measure was the Hp eradication rate at 4-6 weeks after completion of treatment which was confirmed by a negative of 13 UBT. Secondary outcome measures included side effects, impact factor and changes of microbiome after the therapy.

ELIGIBILITY:
Inclusion Criteria:

* children 6-18 years of age who were referred for upper endoscopy and confirmed to have Hp infection

Exclusion Criteria:

* patients were excluded if they had taken proton pump inhibitors, H2-receptor antagonists or antibiotics in the 4 weeks prior to the study. Patients with known antibiotic allergy,hepatic impairment or kidney failure were also excluded. Patients who received Hp therapy before were also excluded.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1440 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
13C-UBT | 13C-UBT was assessed at 4-6 weeks after completion of therapy
  13C-UBT was used to determine whether Hp treatments was successful

SECONDARY OUTCOMES:
side effects | assess at 2,4-6weeks after completion of the therapy
  such as diarrea,rash,dark stool
changes of Shannon diversity indices for gut microbiome | assess at 0,2,4-6weeks after completion of the therapy
  changes of the Shannon diversity indices
changes of OTU for gut microbiome | assess at 0,2,4-6weeks after completion of the therapy
  changes of OTU
changes of abundances for gut microbiome | assess at ,2,4-6weeks after completion of the therapy
  changes of abundances of the bacteria
CYP2C19 gene that impact the metabolism of PPI | detect the gene before the therapy
  CYP2C19 gene polymorphism
virulence gene-cagA | detect the gene before the therapy
  cagA
virulence gene-vacA | detect the gene before the therapy
  vacA
patient compliance | assess compliance 2 weeks after the therapy
  good compliance is defined as taking more than 80% drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones NL, Koletzko S, Goodman K, Bontems P, Cadranel S, Casswall T, Czinn S, Gold BD, Guarner J, Elitsur Y, Homan M, Kalach N, Kori M, Madrazo A, Megraud F, Papadopoulou A, Rowland M; ESPGHAN, NASPGHAN. Joint ESPGHAN/NASPGHAN Guidelines for the Management of Helicobacter pylori in Children and Adolescents (Update 2016). J Pediatr Gastroenterol Nutr. 2017 Jun;64(6):991-1003. doi: 10.1097/MPG.0000000000001594. PMID 28541262

DOCUMENTS (2):
  • Study Protocol (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03365609/Prot_001.pdf
  • Informed Consent Form (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03365609/ICF_000.pdf